CLINICAL TRIAL: NCT01264510
Title: The Evaluation of the Effectiveness of Bone-anchored Hearing Aids (Baha) in Patients With Conductive or Mixed Hearing Loss, or Unilateral Deafness
Brief Title: Evaluation of the Effectiveness of Bone-anchored Hearing Aids (Baha)
Acronym: Baha
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: reason unknown
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/074
Record Dates: First submitted 2010-04-22; First posted 2010-12-21 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Conductive Hearing Loss; Mixed Hearing Loss; Unilateral Deafness
Keywords: conductive hearing loss; mixed hearing loss; unilateral deafness; implanted with Baha; conductive or mixed hearing loss implanted with a Baha or; unilateral deafness implanted with a Baha
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Hearing Loss, Unilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients implanted with a Bone-anchored hearing aid(Baha) (Other)
  Interventions: Other: audiological test battery

INTERVENTIONS:
Other: audiological test battery — routine audiological measurements.

SUMMARY:
A bone-anchored hearing aid (Baha) consists of a titanium implant located at the mastoid, and a sound processor connected with the implant. The sound processor delivers bone conducted stimuli to the cochlea, bypassing the outer and middle ear.

Some patients who are unable to wear or do not benefit from a conventional air-conduction hearing aid, are candidate for a Baha. Typically, these patients suffer from a conductive or a mixed hearing loss. Recently however, Baha's are also being recommended in patients with unilateral deafness. Sound coming from the deaf side is captured and transmitted through bone conduction to the normal inner ear. The overall benefit of a Baha is more difficult to assess in those patients.

Therefore, the goal of the current study is to examine the benefit of a Baha in patients with different audiological profiles (unilateral or bilateral conductive or mixed hearing loss, and unilateral deafness). Special attention will be given to predictive determinants of the benefit with a Baha, and to the improvement of pre-operative criteria and counseling of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients (males and females) already implanted with a bone-anchored hearing aid (Baha) are included in the study.
* Only patients above 18 years will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
benefit of a Bone-anchored hearing aid (Baha) in patients with different audiological profiles | after 3 months up to 10 years
  Patients who are already implanted with a Baha at the University Hospital of Ghent will be re-evaluated once using an audiological test battery. This evaluation will take place at least 3 months after implantation for the recently implanted subjects. For the subjects who are implanted in the past, this evaluation will take place maximum 10 years after implantation. The audiological test battery includes measurements of hearing thresholds, speech understanding in quiet and noise, and auditory orientation tests.

SECONDARY OUTCOMES:
evaluation of subjective benefit of the Baha | after 3 months
  The subjective benefit of the Baha in different situations will be evaluated by means of questionnaires. No measures regarding safety, tolerability or pain will be evaluated because these measures are already verified for the Baha. The outcome measures are strictly related to audiological factors (e.g. the difference in hearing thresholds/ speech understanding/ orientation with and without Baha). The test duration is estimated at 2 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Dhooge, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent — http://www.uzgent.be